CLINICAL TRIAL: NCT04565977
Title: Evaluating Off-label Use of Direct Oral Anticoagulants (DOACs) in Hypercoagulable States
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 042.PHA.2020.A
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Hypercoagulable States
MeSH Terms: conditions — Thrombophilia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Retrospective Cohort: All patients with hypercoagulable states identified by ICD-9/ICD-10 codes from January 1st, 2015 to December 31st, 2019
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Retrospective chart review

SUMMARY:
Retrospective, cohort study chart review in patients with hypercoagulable states.

DETAILED DESCRIPTION:
* Retrospective, cohort study chart review in patients at Methodist Health System
* Data will be pulled on all patients with hypercoagulable states identified by ICD-9/ICD-10 codes from January 1st, 2015 to December 31st, 2019

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 year-old
* Patients with diagnosis of hypercoagulable state identified by ICD-9/ICD-10 codes
* Patients who were prescribed DOACs or VKA for primary or secondary prevention of thrombosis

Exclusion Criteria:

* Patients with FDA-approved indications of oral anticoagulants including atrial fibrillation or treatment/prevention of thrombotic events unrelated to specified hypercoagulable states
* Patients with incomplete electronic medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypercoagulable states identified by ICD-9/ICD-10 codes from January 1st, 2015 to December 31st, 2019
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Rates of thrombotic events during the study period | Jan 1,2015 - Dec 31st, 2019
  Rates of thrombotic events during the study period
Rates of hemorrhagic events during the study period | Jan 1,2015 - Dec 31st, 2019
  Rates of hemorrhagic events during the study period

SECONDARY OUTCOMES:
Rates of DOAC prescribing for thrombosis prevention in hypercoagulable states | Jan 1,2015 - Dec 31st, 2019
  Rates of DOAC prescribing for thrombosis prevention in hypercoagulable states

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Vuylsteke, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No